CLINICAL TRIAL: NCT06934564
Title: De-Implementation of Low-value Testing in Patients Undergoing Low-Risk Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Lesly Ann Dossett, Research Professor of Cancer Quality Improvement, University of Michigan
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00261786; R01HS029306 (AHRQ)
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Breast Lumpectomy; Laparoscopic Cholecystectomy; Inguinal Hernia Repair
Keywords: Preoperative testing

STUDY DESIGN:
Intervention Model Description: Using a stepped wedge design, sixteen Michigan Value Collaborative (MVC)/Michigan Surgical Quality Collaborative (MSQC) sites in Michigan will implement a multi-level, multi-component de-implementation strategy and collect information on the use of unnecessary preoperative testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Wave 1 (Experimental): Each wave will include usual care, preparation (8 weeks before intervention), active de-implementation interventions, and sustainment phases.
  Intervention is Year 1 Quarter 2
  Interventions: Behavioral: Active de-Implementation
- Wave 2 (Experimental): Each wave will include usual care, preparation (8 weeks before intervention), active de-implementation interventions, and sustainment phases.
  Intervention is Year 1 Quarter 3
  Interventions: Behavioral: Active de-Implementation
- Wave 3 (Experimental): Each wave will include usual care, preparation (8 weeks before intervention), active de-implementation interventions, and sustainment phases.
  Intervention is Year 1 Quarter 4
  Interventions: Behavioral: Active de-Implementation
- Wave 4 (Experimental): Each wave will include usual care, preparation (8 weeks before intervention), active de-implementation interventions, and sustainment phases.
  Intervention is Year 2 Quarter 1
  Interventions: Behavioral: Active de-Implementation
- Wave 5 (Experimental): Each wave will include usual care, preparation (8 weeks before intervention), active de-implementation interventions, and sustainment phases.
  Intervention is Year 2 Quarter 2
  Interventions: Behavioral: Active de-Implementation
- Wave 6 (Experimental): Each wave will include usual care, preparation (8 weeks before intervention), active de-implementation interventions, and sustainment phases.
  Intervention is Year 2 Quarter 3
  Interventions: Behavioral: Active de-Implementation

INTERVENTIONS:
Behavioral: Active de-Implementation — During active de-implementation (3 months), the local team will distribute the strategy components (i.e., clinician education, decision support, evaluation, consensus building around perioperative testing pathways, facility-specific feedback, and a pay-for-performance incentive) at the local site.

SUMMARY:
This trial aims to evaluate the effectiveness of a multi-level, multi-component de-implementation strategy to reduce unnecessary preoperative testing. Sixteen Michigan Value Collaborative (MVC)/Michigan Surgical Quality Collaborative (MSQC) sites in Michigan will implement several tools that have been proven to reduce unnecessary testing at a single site, including clinician education, a decision aid, audit and feedback on performance, and a pay-for-performance incentive. The researchers believe that, through the use of these strategies, there will be a significant reduction in unnecessary preoperative testing during the intervention.

ELIGIBILITY:
Site

Inclusion Criteria:

* Over 30% of testing rates on at least one of the three index procedures (breast lumpectomy, laparoscopic cholecystectomy, and inguinal hernia repair)

Exclusion Criteria:

* none

Surgical participants must be over 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of tests within 30 days of surgery not associated with an emergency department visit | Within 30 days of surgery
  Only tests relating to three index procedures; breast lumpectomy, laparoscopic cholecystectomy, and inguinal hernia repair
  Data collected using MVC/MSQC database

SECONDARY OUTCOMES:
Number of unnecessary preoperative testing before low-risk surgery at MVC/MSQC sites not participating in the trial | Up to year 2, quarter 4
  Example related operations: laparoscopic hysterectomy, knee arthroscopy
30-day episode-based spending | Up to Year 2, Quarter 2
  Using the MVC claims data for total spending amounts
Number of unnecessary preoperative testing before low-risk surgery at trial sites | Up to year 2, quarter 4
  Example related operations: laparoscopic hysterectomy, knee arthroscopy
Number of intraoperative complications | Up to year 2, quarter 4
  Examples: myocardial infarction, stroke
Number of same-day case cancellations | Up to year 2, quarter 4

CONTACTS AND LOCATIONS:
Overall Officials: Lesly Dossett, MD, MPH, Principal Investigator — University of Michigan; Hari Nathan, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan and other Michigan Surgical Quality Collaborative sites, Ann Arbor, Michigan, United States